CLINICAL TRIAL: NCT02572128
Title: Comparative Evaluations of Micronutrient Absorption From Mineral Fortified Rice Produced With Different Fortification Techniques: An Evaluation of Hot and Cold Extrusion (Study 1) and Coating Technologies (Study 2)
Brief Title: Mineral Absorption From Fortified Rice Produced With Different Fortification Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); Global Alliance for Improved Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Rice_FeZnEC
Record Dates: First submitted 2015-04-15; First posted 2015-10-08 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study 1 (Experimental): Iron fortified rice hot or cold extruded.
  Interventions: Other: Fortified rice
- Study 2 (Experimental): Iron and zinc fortified rice hot extruded or coated.
  Interventions: Other: Fortified rice

INTERVENTIONS:
Other: Fortified rice — Study 1: Hot or cold extruded rice fortified test meals fortified with Ferric Pyrophosphate and Zinc oxide will be administered - subjects serve as their own controls.
  Study 2: Hot extruded rice or coated rice fortified with Ferric Pyrophosphate and Zinc Oxide will be administered.
  Regular rice fortified with Ferrous Sulfate (FeSO4) will act as a control in study 2.

SUMMARY:
The investigators studies will compare iron, respectively iron and zinc bioavailability from fortified rice produced from different fortification techniques using stable isotopic labels. Study 1 aims to compare the iron bioavailability from hot and cold extruded rice, in Study 2 the iron and zinc bioavailability from rice using one coating technique and hot extrusion will be compared.

DETAILED DESCRIPTION:
Both studies will have a randomized single-blind, cross-over design. Study 1 will be conducted at the Institute for Nutrition and Health (IFNH), Swiss Federal Institute of Technology (ETH) Zurich exclusively; Study 2 will be conducted partly at Clinical Trials Center (CTC) Zurich and at Institute for Nutrition and Health (IFNH).

Study 1: From an initial screening of interested candidates, the investigators will include 20 participants to participate in the study. The participants will consume two different test meals containing 48g regular Basmati rice and 2g fortified rice with a vegetable sauce (in a random order as defined in the study plan). The meals will be based on fortified rice fortified with 57FePP, ZnO and a micronutrient mix, produced with hot (meal A) or cold (meal B) extrusion. The micronutrient mix will contain per served meal 170 µg Folic acid, 1.3 µg vitamin B12, 0.195 mg Vitamin A, 0.65 mg thiamin, 9.1 mg niacin, 0.78 mg vitamin B6 (17) as well as 1,26 mg citric acid and 36,16 mg trisodium-citrate serving as an enhancer for iron absorption. Randomization will include the random order of test meal A and B. Stable iron isotopes will be incorporated in the fortified rice.

The whole study duration from the screening to the last contact with the participant will be about 1 month (36 days, including screening). At screening, on the days of test meal administration and at the study endpoint visit, the participants will spend about 30 minutes at the IFNH in the morning (0700 - 0900h).

Study 2: From an initial screening of interested candidates, 24 non-pregnant non-lactating women will be recruited. The participants will be randomly assigned to one of 3 cohorts (1, 2, 3). The only differences between the cohorts will be the time of study-start and the time of reference meal administration. The participants will consume two different test meals (in a random order as defined in the study plan) and one reference meal. The meals will be based on rice fortified with stable isotopes of iron (57FePP) and zinc (67ZnO) as well as a micronutrient mix, produced with coated rice from Wright Enrichment Inc. (meal A) or hot extruded rice produced at ETH Zurich (meal B). The reference meal (meal C) will consist of extruded rice with the micronutrient mix only (with no extra added iron or zinc) and regular rice where a 58FeSO4 (Ferrous Sulfate) solution is added prior to consumption. Randomization will include the random order of test meals A and B. Meal C will be given one day before the first (cohort 1) or second (cohort 2) test meal. Additionally, stable zinc isotopes will be given to the subjects intravenously.

The whole study duration from the screening to the last contact with the participant will be about 2 months (51 days including screening). At screening and on the days of test meal administration, the participants will spend about 20 - 30 minutes at the IFNH or at the CTC in the morning (0700 - 0900h).

For both studies, the blood samples will be used for determining iron bioavailability. In Study 2, additional urine samples will be collected for determining the zinc bioavailability. The baseline blood and urine samples and the blood samples collected 14 days (Study 1), respectively 15 days (Study 2), after test meal administration as well as the urine samples collected 4 days (96 hours) after test meal administration will be analyzed by inductively coupled plasma mass spectrometry (ICP-MS) for isotope enrichment, and fractional as well as absolute Fe and Zn absorption will be calculated for each test meal in each subject.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* Normal body Mass Index (18.5 - 25 kg/m2)
* Body weight < 65 kg
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by a pregnancy test) or intention to become pregnant during the study
* Lactating/ Breastfeeding
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration and during the intervention time
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months and during the intervention time
* Earlier participation in a study using Fe or Zn stable isotopes or participation in any clinical study within the last 30 days
* Participants who cannot be expected to comply with the study protocol (e.g. not available on certain study appointments)
* Smoking
* Vegan diet

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Study 1: Fractional iron absorption; | 6 months
  Fractional iron (Study 1 and 2) absorption from different isotopically labelled meals will be calculated based on the shift of the isotope ratios in collected blood (for iron determination) samples. The iron absorption will be assessed from blood samples collected 14 or 15 days after meal administration. Iron isotope ratios will be determined by mass spectrometry. Total absorbed iron: measurement unit = mg; Fractional absorbed zinc: measurement unit = %
Study 2: Additionally fractional Zinc absorption | 3 months
  Fractional zinc (Study 2) absorption from different isotopically labelled meals will be calculated based on the shift of the isotope ratios in collected urine (for zinc determination) samples. The zinc absorption will be assessed from urine samples collected 4 days after meal administration. Zinc isotope ratios will be determined by mass spectrometry. Total absorbed zinc: measurement unit = mg; Fractional absorbed zinc: measurement unit = %

SECONDARY OUTCOMES:
Hemoglobin | 6 months
  The secondary outcomes in both studies are the assessment of haemoglobin, plasma ferritin and c-reactive protein in the participants. Unit: mg/l
Plasma Ferritin | 6 months
  The secondary outcomes in both studies are the assessment of haemoglobin, plasma ferritin and c-reactive protein in the participants. Unit: mg/l
C- Reactive Protein | 6 months
  The secondary outcomes in both studies are the assessment of haemoglobin, plasma ferritin and c-reactive protein in the participants. Unit: mg/l
Plasma Zinc | 6 months
  This secondary outcome will be assessed in study 2 only. Unit: mg/l

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof. Dr., Principal Investigator — Head of Laboratory
Locations (2):
- Switzerland (2):
  - Clinical Trials Center, University Hospital, Zurich, Canton of Zurich
  - Human Nutrition Laboratory, ETH Zurich, Zurich